CLINICAL TRIAL: NCT01883583
Title: Pilot Study of Contrast-Enhanced Ultrasound of Transplanted Kidney for Evaluation of Effectiveness of Perfusion Parameter in Assessment of Allograft Nephropathy
Brief Title: Pilot Study of Contrast-Enhanced Ultrasound of Transplanted Kidney
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Yeon Cho, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SeoulNUH-rad2
Record Dates: First submitted 2013-06-15; First posted 2013-06-21 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Transplant; Failure, Kidney
Keywords: Ultrasound; Perfusion Imaging; Elasticity Imaging Techniques; Kidney Transplantation; Graft Rejection; Chronic allograft nephropathy
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pilot group (Experimental): Contrast-enhanced Ultrasound And Sonoelastography of transplanted kidney will be performed for acquisition of a number of parameters and time-intensity curves, before ultrasound guided biopsy of transplanted kidney.
  Interventions: Device: Contrast-enhanced Ultrasound And Sonoelastography

INTERVENTIONS:
Device: Contrast-enhanced Ultrasound And Sonoelastography — Before ultrasound guided biopsy of transplanted kidney, we will perform conventional, Sonoelastography and real-time contrast-enhanced ultrasound using Sonovue for acquisition of parameters and data, respectively.

SUMMARY:
To check the possibility of the acquisition of a number of parameters through real-time contrast-enhanced ultrasound and sonoelastography images and to verify the correlation with pathologic results from ultrasound guided biopsy of transplanted kidney

DETAILED DESCRIPTION:
To check the possibility of the acquisition of a number of parameters through real-time contrast-enhanced ultrasound and sonoelastography images and to verify the correlation with pathologic results from ultrasound guided biopsy of transplanted kidney.

Ten patients scheduled to perform ultrasound guided biopsy of transplanted kidney will be enrolled. The patients who have previous medical history of cardiac problem or who do not recover renal function over three days after graft surgery will be excluded.

Before ultrasound guided biopsy of transplanted kidney, we will perform conventional, Sonoelastography and real-time contrast-enhanced ultrasound using Sonovue for acquisition of parameters and data, respectively. We will check the possibility of the acquisition of a number of parameters through real-time contrast-enhanced ultrasound and sonoelastography images using analyzing program (VueBox, Bracco, Swiss). And we will verify the correlation of acquired data and parameters with pathologic results from ultrasound guided biopsy of transplanted kidney.

From perfusion images, several regions of interest (ROIs) will be marked including main renal artery, segmental artery and renal medulla. A number of time-intensity curves (TICs) are acquired from ROIs using VueBox.

The parameters acquired from time intensity curve (TIC) (i.e. arrival time, mean transit time, time to peak, basal intensity, peak intensity, area under curve, slope rate of ascending and descending curves), the date acquired from spectral Doppler ultrasound (i.e. restive index, pulsatility index) and Values of shear wave velocities of the several regions of interest acquired from Sonoelastography will be analyzed to find statistical significance in assessment of allograft nephropathy such as acute rejection or chronic allograft nephropathy.

Pathologic conditions such as acute rejection may show the decrease in arrival time, peak intensity, area under curve suggesting total blood flow and accelerating slope rate, compared with non-pathologic condition.

ELIGIBILITY:
Inclusion Criteria:

* 1)Patients to perform ultrasound guided biopsy of transplanted kidney

Exclusion Criteria:

* 1)Patients to have the medical histories of heart such as acute failure, arrhythmia, ischemia, infarction and angioplasty 2)Patients to show poor graft function which does not recovery within three days after transplantation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Acquisition of time-intensity curve(TIC) using contrast-enhanced ultrasound | The day of admission (within 24hours)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Yeon Cho, Professor, Principal Investigator — Department of Radiology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea